CLINICAL TRIAL: NCT01450800
Title: Antibiotic Prophylaxis for Urinary Tract Infection in Patients Requiring Catheterization After Urogynecologic Surgery
Brief Title: Suppressive Therapy With Oral Antibiotics for Prevention of Postoperative Urinary Tract Infection (UTI)
Acronym: STOPP UTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00025269; 3913577 (Other Grant/Funding Number: Charles B Hammond Research Fund)
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Urinary Tract Infection
Keywords: urinary tract infection; gynecologic surgery; post-operative complications; nitrofurantoin
MeSH Terms: conditions — Urinary Tract Infections | interventions — Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrofurantoin (Active Comparator): Nitrofurantoin 100mg by mouth daily starting on postoperative day 1 for up to 7 days during catheterization
  Interventions: Drug: Nitrofurantoin
- Placebo (Placebo Comparator): Placebo drug 1 tablet by mouth daily starting on postoperative day 1 for up to 7 days during catheterization
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrofurantoin — Nitrofurantoin 100mg po daily to be taken every day the patient uses a catheter for up to one week post-operatively
  Other Names: Macrobid; Macrodantin
  Arms: Nitrofurantoin
Drug: Placebo — Participants randomized to placebo will be instructed to take placebo one tablet by mouth daily starting on postoperative day 1 for up to 7 days during catheterization
  Other Names: Placebo medication; Inactive medication
  Arms: Placebo

SUMMARY:
This is a study of patients undergoing gynecologic surgery who require post-operative catheterization to determine if prophylactic antibiotic treatment decreases the risk of post-operative urinary tract infection in these patients.

DETAILED DESCRIPTION:
Study Population Participants will be recruited from all patients who are planning to undergo gynecologic surgery by an attending surgeon in the Division of Urogynecology at Duke University Medical Center (DUMC). After enrollment and randomization, the participants will take the study drug once daily to start on post-operative day one and continue until the participant has stopped catheterizing for up to one week after surgery. The participant will also complete a daily diary for one week after surgery to record any catheterization and any study drug or additional antibiotic medication taken. We will then follow patients for a total of three weeks after surgery to monitor for treatment for UTI. At three weeks after surgery the observation period for the participant is complete.

Sample Size Under the assumption of 80% power and an alpha error of 0.05, we would need 156 subjects to demonstrate a 66% reduction in risk of UTI (i.e. from 28% to 10%) in those undergoing prophylactic antibiotic treatment. Therefore, we aim to recruit a total of 175 participants to account for participant dropout.

Study Definitions For our study purposes, post-operative catheterization will be defined to include patients who are hospitalized post-operatively with an indwelling Foley catheter as well as patients discharged with either intermittent self-catheterization (ISC) or indwelling Foley catheter. The decision to catheterize will be determined by type of surgical procedure, need for inpatient stay and void trial results. Void trials will be conducted as follows: the bladder is backfilled with 300cc normal saline, the catheter is removed and the patient is prompted to void immediately and, after voiding is complete, a (PVR) post-void residual volume is measured. The patient passes the void trial if she voids over 200cc in total volume or if her PVR is less than 100cc.

Our primary outcome of treatment for UTI within the first three weeks after surgery is to be defined clinically. A patient will be considered to have received treatment for UTI if she receives any antibiotic therapy for clinically suspected or culture-proven urinary tract infection (i.e. empirically given upon development of urinary symptoms or prescribed based on urinalysis or urine culture results) within the first three weeks after surgery.

Data Collection Demographic characteristics, operative data and post-operative data will be collected. Prior to discharge after surgery all patients will undergo a void trial per standard procedure unless they receive an indwelling Foley catheter for overnight hospitalization. Post-operatively all subjects will be given a catheterization diary to record days of catheterization and days of antibiotic therapy. All subjects will be instructed to call our clinical office to report any urinary complaints and/or treatment for UTI. Information will be collected from electronic medical records regarding any office visits, urine cultures performed or treatment for UTI during this post-operative period. Data will be entered into a de-identified study database for analysis by the PI and study coordinator who will be blinded to participant randomization.

Subject Randomization and Blinding Study participants will be randomized to prophylactic treatment versus no treatment via a computerized randomization scheme by the IDS at the time of enrollment. Patients will be blinded to treatment by the utilization of placebo tablets.

Adverse Events Nitrofurantoin is FDA approved for the treatment of UTI. We will be using a prophylactic dose and will monitor for any adverse events. Adverse events will be reported per protocol. A safety monitoring designee will perform reviews on a designated basis throughout the study.

Study Costs There will be no additional cost to the patient for their participation in this study. No additional laboratory testing will be performed as a result of participation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing urogynecologic surgery
* Receive postoperative catheterization

Exclusion Criteria:

* Age less than 21 years old
* Pregnancy
* Allergy, contraindication or intolerance to Nitrofurantoin
* Do not speak English
* Dependent on trans-urethral catheter to accomplish voiding preoperatively
* Undergoing interstim device placement, urethral diverticulum surgery or fistula surgery
* Sustain intraoperative urinary tract injury requiring postoperative catheterization

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Amundsen, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Brown JS, Grady D, Ouslander JG, Herzog AR, Varner RE, Posner SF. Prevalence of urinary incontinence and associated risk factors in postmenopausal women. Heart & Estrogen/Progestin Replacement Study (HERS) Research Group. Obstet Gynecol. 1999 Jul;94(1):66-70. doi: 10.1016/s0029-7844(99)00263-x. PMID 10389720
- [Background] Hannestad YS, Rortveit G, Sandvik H, Hunskaar S; Norwegian EPINCONT study. Epidemiology of Incontinence in the County of Nord-Trondelag. A community-based epidemiological survey of female urinary incontinence: the Norwegian EPINCONT study. Epidemiology of Incontinence in the County of Nord-Trondelag. J Clin Epidemiol. 2000 Nov;53(11):1150-7. doi: 10.1016/s0895-4356(00)00232-8. PMID 11106889
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Thomas TM, Plymat KR, Blannin J, Meade TW. Prevalence of urinary incontinence. Br Med J. 1980 Nov 8;281(6250):1243-5. doi: 10.1136/bmj.281.6250.1243. PMID 7427654
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Levin I, Groutz A, Gold R, Pauzner D, Lessing JB, Gordon D. Surgical complications and medium-term outcome results of tension-free vaginal tape: a prospective study of 313 consecutive patients. Neurourol Urodyn. 2004;23(1):7-9. doi: 10.1002/nau.10164. PMID 14694449
- [Background] Nilsson CG, Kuuva N, Falconer C, Rezapour M, Ulmsten U. Long-term results of the tension-free vaginal tape (TVT) procedure for surgical treatment of female stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12 Suppl 2:S5-8. doi: 10.1007/s001920170003. PMID 11450979
- [Background] Falagas ME, Athanasiou S, Iavazzo C, Tokas T, Antsaklis A. Urinary tract infections after pelvic floor gynecological surgery: prevalence and effect of antimicrobial prophylaxis. A systematic review. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1165-72. doi: 10.1007/s00192-008-0584-0. Epub 2008 Apr 10. PMID 18401538
- [Background] Sutkin G, Lowder JL, Smith KJ. Prophylactic antibiotics to prevent urinary tract infection during clean intermittent self-catheterization (CISC) for management of voiding dysfunction after prolapse and incontinence surgery: a decision analysis. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Aug;20(8):933-8. doi: 10.1007/s00192-009-0885-y. Epub 2009 Apr 10. PMID 19582384
- [Background] Macy E, Poon K-Y T. Self-reported antibiotic allergy incidence and prevalence: age and sex effects. Am J Med. 2009 Aug;122(8):778.e1-7. doi: 10.1016/j.amjmed.2009.01.034. PMID 19635279
- [Derived] Dieter AA, Amundsen CL, Edenfield AL, Kawasaki A, Levin PJ, Visco AG, Siddiqui NY. Oral antibiotics to prevent postoperative urinary tract infection: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):96-103. doi: 10.1097/AOG.0000000000000024. PMID 24463669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who received postoperative transurethral catheterization after surgery for pelvic organ prolapse, urinary incontinence, or both by the Division of Urogynecology at Duke University Medical Center from 8/2011 through 2/2013 were identified, recruited and enrolled after providing written informed consent at a routine pre-operative visit.
Pre-assignment Details: Randomization occurred within a few hours after surgery. Participants were excluded prior to randomization if they sustained intraoperative injury to the urinary tract requiring prolonged catheterization, or if they passed an immediate void trial on day of surgery (as these participants did not receive additional postoperative catheterization).
Groups:
- Nitrofurantoin: Randomized to nitrofurantoin 100mg daily for each day of catheterization for up to 7 days
- Placebo: Randomized to placebo 1 tablet daily for each day of catheterization for up to 7 days
Period: Overall Study
Arm/Group | Nitrofurantoin | Placebo
Started | 82 (82 participants were randomized to nitrofurantoin) | 81 (81 participants were randomized to placebo)
Completed | 81 | 78
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Population: 163 participants were randomized, 82 to nitrofurantoin and 81 to placebo. Four randomized participants were excluded from the final analysis. One in the placebo group was excluded, as she had previously been included in the study during a prior surgery. Three participants in the nitrofurantoin group were excluded due to protocol deviations.
Groups:
- Nitrofurantoin: Participants randomized to receive antibiotics instructed to take nitrofurantoin 100mg by mouth daily starting on postoperative day 1 for up to 7 days during catheterization
- Placebo: Participants randomized to receive placebo instructed to take placebo 1 tablet by mouth daily starting on postoperative day 1 for up to 7 days during catheterization
- Total: Total of all reporting groups
Arm/Group | Nitrofurantoin | Placebo | Total
Number analyzed (Participants) | 82 | 81 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 55 | 113
  >=65 years | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 57 (13) | 57 (13)
Gender [Count of Participants; unit: Participants]
  Female | 82 | 81 | 163
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 82 | 81 | 163

OUTCOME MEASURES:

1. Primary Outcome: Urinary Tract Infections
Description: The primary outcome was treatment for UTI within the first 3 weeks after surgery. Treatment for UTI was defined to include any treatment received for clinically suspected or culture-proven urinary tract infection within 3 weeks of surgery. Clinically suspected treatment was defined to include treatment given empirically upon development of urinary symptoms or prescribed based on urine test results. Culture-proven UTI was defined as a urine culture with greater than 100,000 colony-forming units of a single organism.
Time Frame: three weeks post-operative
Population: Intent-to-treat analysis
Measure: Number; unit: participants
Groups:
- Nitrofurantoin: Randomized to nitrofurantoin 100mg daily while using a catheter for up to 7 days
- Placebo: Randomized to placebo 1 tab daily while using a catheter for up to 7 days
Arm/Group | Nitrofurantoin | Placebo
Number analyzed (Participants) | 81 | 78
participants | 18 | 10

2. Secondary Outcome: Other Risk Factors for UTI
Description: We examined risk of UTI as related to vaginal estrogen therapy
Time Frame: 3 weeks following surgery
Population: Used entire study population to determine risk factors for UTI
Measure: Number; unit: participants
Groups:
- All Participants in Final Analysis: All participants in the final analysis were examined
Arm/Group | All Participants in Final Analysis
Number analyzed (Participants) | 159
participants
  participants with no UTI | 131
  participants with UTI not on vaginal estrogen | 24
  participants with UTI on vaginal estrogen | 4

3. Secondary Outcome: Other Risk Factors for UTI
Description: We examined risk of UTI as related to history of recurrent UTIs
Time Frame: 3 weeks following surgery
Population: Used entire study population to determine risk factors for UTI
Measure: Number; unit: participants
Arm/Group | All Participants in Final Analysis
Number analyzed (Participants) | 159
participants
  participants with no UTI | 131
  participants with UTI with recurrent UTI | 4
  participants with UTI with no recurrent UTI | 24

4. Secondary Outcome: Other Risk Factors for UTI
Description: We examined risk of UTI as related to preoperative UTI treatment
Time Frame: 3 weeks following surgery
Population: Used entire study population to determine risk factors for UTI
Measure: Number; unit: participants
Arm/Group | All Participants in Final Analysis
Number analyzed (Participants) | 159
participants
  participants without UTI | 131
  participants with UTI with preoperative UTI | 3
  participants with UTI with no preoperative UTI | 25

5. Secondary Outcome: Other Risk Factors for UTI
Description: We examined risk of UTI as related to Creatinine Clearance
Time Frame: 3 weeks following surgery
Population: Used entire study population to determine risk factors for UTI
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | All Participants in Final Analysis
Number analyzed (Participants) | 159
mL/min
  Participants with UTI | 115 (37)
  Participants without UTI | 101 (30)

6. Secondary Outcome: Other Risk Factors for UTI
Description: We examined risk of UTI as related to sling as part of surgery
Time Frame: 3 weeks following surgery
Population: Used entire study population to determine risk factors for UTI
Measure: Number; unit: participants
Arm/Group | All Participants in Final Analysis
Number analyzed (Participants) | 159
participants
  participants with no UTI | 131
  participants with UTI with sling | 16
  participants with UTI with no sling | 12

7. Secondary Outcome: Other Risk Factors for UTI
Description: We examined risk of UTI as related to total postoperative catheter days
Time Frame: 3 weeks following surgery
Population: Used entire study population to determine risk factors for UTI
Measure: Median (95% Confidence Interval); unit: days of catheterization
Arm/Group | All Participants in Final Analysis
Number analyzed (Participants) | 159
days of catheterization
  Participants with UTI | 2 [1 to 4]
  participants without UTI | 1 [1 to 3]

8. Secondary Outcome: Other Risk Factors for UTI
Description: We examined risk of UTI as related to postoperative catheter type
Time Frame: 3 weeks following surgery
Population: Used entire study population to determine risk factors for UTI
Measure: Number; unit: participants
Arm/Group | All Participants in Final Analysis
Number analyzed (Participants) | 159
participants
  participants without UTI | 131
  participants with UTI with Foley | 25
  participants with UTI with self-catheterization | 3

9. Other Pre Specified Outcome: Antibiotic Resistance to Macrobid
Description: We examined for macrobid resistance on urine culture results within 3 weeks of surgery
Time Frame: 6 weeks after surgery
Population: Examined urine cultures with susceptibility testing results for all participants who had positive urine culture results
Measure: Number; unit: urine culture resistant to nitrofurantoi
Groups:
- Urine Cultures Performed: All participants in the final analysis were examined
Arm/Group | Urine Cultures Performed
Number analyzed (Participants) | 9
urine culture resistant to nitrofurantoi | 1

ADVERSE EVENTS:
Time Frame: 20 months
Groups:
- Nitrofurantoin: Participants randomized to receive nitrofurantoin 100mg by mouth daily each day of catheterization for up to one week after surgery
- Placebo: Participants randomized to receive placebo 1 tablet by mouth daily each day of catheterization for up to one week after surgery
Arm/Group | Nitrofurantoin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81

LIMITATIONS AND CAVEATS:
Limitations of our study include recall bias and selection bias. Our findings have limited applicability to elderly patients undergoing pelvic reconstructive surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes